CLINICAL TRIAL: NCT06166082
Title: Stanford Neuromodulation Therapy (SNT) for the Treatment-Resistant Depression: A Study Multicenter, Randomized, Double-blind, Placebo Parallel Controlled Trial
Brief Title: Stanford Neuromodulation Therapy (SNT) for the Treatment-Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changping Laboratory (Other)
Collaborators: Xianyue Hospital, Xiamen (Unknown); Hebei Mental Health Center, Baoding (Unknown); HuiLongGuan Hospital, Beijing (Unknown); Wuhan Mental Health Center, Wuhan (Unknown); Zhumadian Second People's Hospital, Zhumadian (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLSNT_Multicenter
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-12

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment Resistant Depression; TRD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active iTBS-DLPFC (Experimental): The active group will receive active iTBS. Treat 10 times a day with 1800 pulses per day for consecutive 5 days, with 50 minutes inter-session intervals.
  Interventions: Device: Active iTBS-DLPFC
- Sham iTBS-DLPFC (Sham Comparator): The sham group will receive sham iTBS. Treat 10 times a day with 1800 pulses per day for consecutive 5 days, with 50 minutes inter-session intervals.
  Interventions: Device: Sham iTBS-DLPFC

INTERVENTIONS:
Device: Active iTBS-DLPFC — Participants will receive 10 sessions per day of 1800 pulses per session, lasting for 5 days.
  Arms: Active iTBS-DLPFC
Device: Sham iTBS-DLPFC — The parameters in the sham arms are the same as the active stimulation groups. Stimulation was delivered by the same device as the active group fitted with a sham coil.
  Arms: Sham iTBS-DLPFC

SUMMARY:
This study is a multicenter, randomized, double-blind, and sham-controlled trial using the identical protocol as the SNT to replicate the antidepressant efficacy of SNT for TRD. Patients will be recruited and randomly assigned (1:1 ratio) to receive active or sham groups from 5 hospitals in China. The interventions will last for 5 days and both groups will be followed up for 8 weeks on the same time schedules. During the intervention and at least the first 4 weeks of post-treatment, participants will keep a stable antidepressant regimen. The individualized SNT target in the left dorsolateral prefrontal cortex (DLPFC) will be generated from 30 minutes of resting-state functional MRI collected at baseline.

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Training (rTMS) is a non-invasive neuromodulation that has been approved by the Food and Drug Administration (FDA) for treating patients with treatment-resistant depression(TRD). In 2022, the US FDA approved a high-dose intervention called Stanford Neuromodulation Therapy (SNT) to achieve rapid relief of patient symptoms in TRD. This therapy involves 10 1800 pulse Intermittent Theta Burst Stimulation (iTBS) interventions per day for consecutive 5 days on the dorsolateral prefrontal cortex (DLPFC), with 50 minutes inter-session intervals. At the end of the SNT intervention, the response rate reached 71.4% (13.3% in the sham group); At the 4th week follow-up after treatment, the response rate was 69.2% (7.1% in the sham group). This therapy has the advantage of quickly taking effect in the treatment of patients with TRD in a short period. However, there are also some limitations with this therapy, such as the need to undergo 10 high-dose interventions with 1800 pulses per day, which takes about 9 hours and may reduce patient compliance with the treatment. In addition, this study is a single-center small sample trial (14 cases with active and 15 cases with sham stimulation). The SNT therapy brings confidence to TRD patients, its efficacy and safety need to be verified in multicenter, randomized, double-blind, placebo-parallel controlled clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of DSM-5(Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) for depression disorder without psychotic symptoms, and currently experiencing a recurrence episode;
* Hamilton Depression Scale (HAMD-17) scores for 17 items ≥ 20 points, and the Montgomery Asberg Depression Rating Scale (MADRS) score is ≥ 20 points;
* hospitalized/outpatient patients aged ≥ 22 and ≤ 65 years old, male or female;
* The Maudsley Staging Method (MSM) assesses patients as at least moderate refractory (MSM score ≥ 7 points);
* Stable use of antidepressants for 4 weeks before randomization, with the type of antidepressant used being selective serotonin reuptake Selective serotonin reuptake inhibitors (SSRIs) or/and serotonin and norepinephrine reuptake Serotonin-norepinephrine reuptake inhibitors (SNRIs), the therapeutic dose is within the dosage range as the drug manual recommended;
* Understand the trial and sign the informed consent form.

Exclusion Criteria:

* Meets DSM-5 diagnostic criteria for other mental disorders, including schizophrenia spectrum disorders, bipolar and related disorders, and psychiatric disorders Developmental disorders, neurocognitive disorders, or depression caused by substances and/or drugs, or other medical problems;
* Individuals with pacemakers, cochlear implants, or other metal objects, as well as any electronic devices implanted in the body, and those with claustrophobia Contraindications for magnetic resonance imaging scans such as fear, and contraindications for rTMS treatment;
* History of epilepsy (presence of at least 2 uninduced seizures more than 24 hours apart, or diagnosis of the epileptic syndrome, or seizures within the past 12 months); Or currently received medications or other treatments that will lower the seizure threshold Syndromes, or seizures within the past 12 months;
* Received TMS treatment before participating in the trial;
* Individuals who have received ECT or phototherapy within three months;
* No response to ECT treatment (>8 times);
* Previously received antidepressant treatment with implanted devices (such as DBS, VNS);
* Concomitant organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumors, etc.) and a history of severe brain injury;
* Complicated with serious heart, liver, kidney diseases, diabetes, and other serious physical diseases, which cause abnormal symptoms and signs of brain nerves, Or physical exhaustion;
* Women of childbearing age who are currently pregnant, breastfeeding, or planning or may become pregnant during the trial period;
* Substance abuse or dependence (including alcohol, drugs, and other psychoactive substances) in the past year;
* First-degree relatives suffer from bipolar disorder;
* High risk of suicide;
* Difficulty in communication to understand or follow instructions, and unable to cooperate with treatment and evaluation;
* Current in clinical trials of other drugs or physical therapies (DBS, ECT, rTMS);
* The researchers believe it is not suitable to participate.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Pretreatment (baseline), 28 days post-treatment
  A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.The MADRS has an overall score range from 0-60, with higher scores corresponding to higher levels of depression.

SECONDARY OUTCOMES:
Change in MADRS | Baseline, Day 5 (Immediate Post-treatment), 7 days Post-treatment, 14 days Post-treatment, 21 days Post-treatment, 56 days Post-treatment]
  A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.The MADRS has an overall score range from 0-60, with higher scores corresponding to higher levels of depression.
Change in the Hamilton Rating Scale for Depression (HAMD-17) | Baseline, Day 5 (Immediate Post-treatment), 7 days Post-treatment, 14 days Post-treatment, 21 days Post-treatment, 28 days Post-treatment, 56 days Post-treatment]
  A provider administered questionnaire used to assess remission and recovery from depression. The HAMD-17 is a 17-item questionnaire to assess depression severity. Each item is scored from 0-4, with higher scores representing increasing depression severity.
Change in the Hamilton Rating Scale for Depression (HAMD-6) Score | Baseline, Day 1, 2, 3, 4 in treatment, Day 5 (Immediate Post-treatment), 7 days Post-treatment, 14 days Post-treatment, 21 days Post-treatment, 28 days Post-treatment, 56 days Post-treatment]
  The Hamilton Depression Rating Scale (HDRS, also known as Ham-D) is the most widely used clinician-administered depression assessment scale.
  The Ham-6 version consists of 6 items assessing for: mood, guilt, general somatic symptoms, work and activities, anxiety and slowness of thought and speech). Each item is scored on a scale of 0 to 4, except for the somatic symptoms item, which is scored 0 to 2. On the HAM-6 there can be a total score of 22. Higher scores represent higher depression severity. Here, we report a count of participants with an overall increase, decrease or no change in total HAM-6 score.
  Participants with an increase in total score (row 3) would signify a worse outcome than participants with a decrease in total score.
Change in Quick Inventory of Depressive Symptomatology Self-Report (QIDS_SR) | Baseline, Day 5 (Immediate Post-treatment), 7 days Post-treatment, 14 days Post-treatment, 21 days Post-treatment, 28 days Post-treatment, 56 days Post-treatment]
  The 16-item QIDS_SR is a widely used self-report instrument covering depressive symptoms incorporating nine Diagnostic and Statistical Manual of Mental Disorder-IV (DSM-IV) diagnostic criteria for major depressive disorders. Each item is scored on a scale of 0 to 4. Higher scores represent higher depression severity.
Safety estimated using YMRS | Baseline, Day 5 (Immediate Post-treatment)
  Young Mania Rating Scale(YMARS) measures mania
cognitive change in Digit Symbol Substitution Test (DSST） | Baseline, Day 5(Immediate Post-treatment)
  Cognitive scores are measured using Chinese brief cognitive test (C-BCT), the DSST equires a subject to match symbols to numbers according to a key located on the top of the page
cognitive change in continuous performance test (CPT） | Baseline, Day 5(Immediate Post-treatment)
  CPT from the C-BCT measures a person's sustained and selective attention
cognitive change in Trail-Making Test (TMT) | Baseline, Day 5(Immediate Post-treatment)
  The TMT test from the C-BCT can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning
cognitive change in Digit Span Test (DST) | Baseline, Day 5(Immediate Post-treatment)
  DST from the C-BCT is a measure of verbal short term and working memory that can be used in two formats, Forward Digit Span and Reverse Digit Span

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (5):
- China (5):
  - Hebei Mental Health Center, Baoding
  - HuiLongGuan Hospital, Beijing
  - Wuhan Mental Health Center, Wuhan
  - Xianyue Hospital, Xiamen
  - Zhumadian Second People's Hospital, Zhumadian